CLINICAL TRIAL: NCT06470958
Title: Investigation of Functional Brain Features in Women with Migraine
Status: Recruiting | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Faisal Mohammad Amin, Principal Investigator, Danish Headache Center
Other Study IDs: H-23054319
Record Dates: First submitted 2024-02-28; First posted 2024-06-24 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Menstrual-related migraine without aura: Migraine patients
- Healthy volunteers: Control group

SUMMARY:
This study aims to investigate whether the functional alterations in the brain of individuals with migraine appear before the peripheral vascular changes. This will be investigated using functional and structural neuroimaging in individuals with spontaneous menstually-related migraine.

DETAILED DESCRIPTION:
Spontaneous migraine attacks are unpredictable and therefore been logistically arduous to investigate in neuroimaging studies. Menstrually-related migraine provides an opportunity to study spontaneous attacks in a controlled imaging setup. The present project aims to investigate women with menstrually-related migraine using daily functional magnetic resonance imaging (MRI) scans 2-3 days before the onset of the menstrual bleeding and until (and including) the headache phase of migraine or up to five consecutive days. A control-group of women without migraine will also be recruited and undergo the same MRI scan protocol.

ELIGIBILITY:
Inclusion Criteria:

For women with migraine

- Episodic menstrually-related migraine without aura > 12 months according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria

For women with migraine and healthy women

* 18-40 years of age
* Weight 50-100 kg
* Regular menstruation

Exclusion Criteria:

For women with migraine

* Other primary headache disorders than migraine, except infrequent episodic tension-type headache according to the ICHD-3 criteria
* Secondary headache disorders
* Headache on the first scan day or 48 hours before the first scan
* Absence of the menstruation for the past 12 months
* Daily intake of medication of any kind except oral contraceptives
* Ingestion of any type of medication later than 4 times the plasma half-life of the substance in question (on the day of the scan), except for oral contraceptives
* Intake of coffee, tea or alcohol 12 hours prior to scan days
* Fertile women not using safe contraception. Fertile women are defined as women without hysterectomy and < 2 years postmenopausal women. Safe contraception includes the intrauterine device, oral contraceptive pills, surgical sterilization of the woman, depot progestogen or condoms
* Change of hormonal contraceptives for the past 3 months
* Perimenstrual syndrome
* Pregnant or breastfeeding women
* Information or clinical signs of:

  * Hypertension (systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg)
  * Low blood pressure (systolic blood pressure < 100 mm Hg and/or diastolic blood pressure < 50 mm Hg)
* Cardiovascular diseases of any kind, including cerebrovascular disease
* Diabetes
* Unregulated mental illness or substance abuse
* Illnesses of any kind deemed incompatible by the examining physician for participation in the study
* Contraindications to MRI (including metal in the body or claustrophobia)
* Do not want to be informed about unexpected pathological findings on the MRI

For healthy women

* History of any primary headache except infrequent episodic tension-type headache according to the ICHD-3 criteria
* First degree family history of primary headache disorders except infrequent episodic tension-type headache according to the ICHD-3 criteria (max five days/month)
* Secondary headache disorders
* Headache during the menstrual period from 2 days before to 2 days after the first menstrual bleeding day
* Headache on the first scan day or 48 hours before the first scan
* Absence of the menstruation for the past 12 months
* Daily intake of medication of any kind except oral contraceptives
* Ingestion of any type of medication later than 4 times the plasma half-life of the substance in question (on the day of the scan), except for oral contraceptives
* Intake of coffee, tea or alcohol 12 hours prior to scan days
* Fertile women not using safe contraception. Fertile women are defined as women without hysterectomy and < 2 years postmenopausal women. Safe contraception includes the intrauterine device, oral contraceptive pills, surgical sterilization of the woman, depot progestogen or condoms
* Change of hormonal contraceptives for the past 3 months
* Pregnant or breastfeeding women
* Perimenstrual syndrome
* Information or clinical signs of:

  * Hypertension (systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg)
  * Low blood pressure (systolic blood pressure <100 mm Hg and/or diastolic blood pressure < 50 mm Hg) Investigation of functional brain features in women with migraine
* Cardiovascular diseases of any kind, including cerebrovascular disease.
* Diabetes
* Unregulated mental illness or substance abuse
* Illnesses of any kind deemed incompatible by the examining physician for participation in the study
* Contraindications to MRI (including metal in the body or claustrophobia)
* Do not want to be informed about unexpected pathological findings on the MRI

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with menstrually-related migraine and women with no history of migraine. All participants have regular menstruation and 18-40 years old.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Brain excitability in migraine patients | Up to 5 days in relation to menstruation
  Changes in the migraine brain excitability in areas related to migraine during the menstrual period. This will be assessed functional magnetic resonance imaging.
Brain connectivity in migraine patients | Up to 5 days in relation to menstruation
  Changes in the migraine brain connectivity in areas related to migraine during the menstrual period. This will be assessed functional magnetic resonance imaging.
Arterial circumference in migraine patients | Up to 5 days in relation to menstruation
  Changes in arterial circumference during the menstrual period. This will assessed using Magnetic Resonance Angiography.
Arterial circumference after rescue medication in migraine patients | Up to 5 days in relation to menstruation
  Changes in arterial circumference after rescue medication in migraine patients. This will assessed using Magnetic Resonance Angiography.
Brain excitability in healthy volunteers | Up to 5 days in relation to menstruation
  Changes in brain excitability or connectivity in areas related to migraine during the menstrual period in healthy volunteers. This will be assessed using functional magnetic resonance imaging.
Brain connectivity in healthy volunteers | Up to 5 days in relation to menstruation
  Changes in brain connectivity in areas related to migraine during the menstrual period in healthy volunteers. This will be assessed using functional magnetic resonance imaging.
Arterial circumference in healthy volunteers | Up to 5 days in relation to menstruation
  Changes in arterial circumference during the menstrual period in healthy volunteers. This will assessed using Magnetic Resonance Angiography.

SECONDARY OUTCOMES:
Migraine attacks during the menstrual period | Up to 7 days in relation to menstruation
  Investigate features of migraine attacks during the menstrual period using a headache questionnaire
Association of the migraine attack features to brain excitability | Up to 5 days in relation to menstruation
  Investigate the association of the migraine attack features to alterations in the brain excitability during the menstrual period. Functional magnetic resonance imaging and headache questionnaire will be used.
Association of the migraine attack features to functional connectivity | Up to 5 days in relation to menstruation
  Investigate the association of the migraine attack features to alterations in the brain functional connectivity during the menstrual period. Functional magnetic resonance imaging and headache questionnaire will be used.
Association of the migraine attack features to vasculature changes | Up to 5 days in relation to menstruation
  Investigate the association of the migraine attack features to alterations in the arterial circumference. Magnetic Resonance Angiography and headache questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Mohammad Amin, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No